CLINICAL TRIAL: NCT04730336
Title: Assessment of the Impact of Tixel Treatment of Periorbital Wrinkles on Dry Eye Symptoms and Signs in Patients With Dry Eye
Brief Title: Assessing the Impact of Tixel Treatment of Periorbital Wrinkles on Dry Eye Symptoms and Signs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UREC 1524
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All participants will undergo three sessions of treatments with the Investigation devise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tixel Treatment (Experimental): Tixel Treatment 3 Tixel treatment sessions, 2 weeks apart follow by 2 Follow up sessions
  Interventions: Device: Tixel

INTERVENTIONS:
Device: Tixel — Peri-Orbital fractional treatment on the Eye-Lid to assess the effect on Dry Eye symptoms
  Other Names: Fractional

SUMMARY:
Pilot study where effect of standard Tixel treatment as used for periorbital wrinkles would be assessed on Dry Eye Disease symptoms and signs

DETAILED DESCRIPTION:
Safety Assessment will be asses via AE/SAE reporting and Impact Assessment of the effect of treatment on dry eye symptoms and signs through multiple test indicate Dry Eye

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mild to Moderate Periorbital wrinkles
* OSDI score of at least 23
* Noninvasive Tear film break up time (NIKBUT) ≤ 10 seconds
* No other eye or skin or immune problems
* Willing and able to provide written informed consent.
* Willing to participate in all study activities and instructions.

Exclusion Criteria:

* Pregnancy and/or breastfeeding
* Lesions in the periorbital area
* Acute severe blepharitis
* Acute conjunctivitis
* Other concomitant anterior eye disease
* Has undergone outdoors/sunbed tanning during the last 4 weeks
* Is unwilling to follow the Tixel aftercare instructions after each of the three Tixel treatments.
* Active Herpes Simplex or tendency for Herpes Simplex in the periorbital area (meaning the subject has had the condition previously).
* Current skin cancer, malignant sites and/or advanced premalignant lesions or moles in the treatment area.
* An impaired immune system condition or use of immunosuppressive medication.
* Collagen disorders, keloid formation and/or abnormal wound healing.
* Previous invasive/ablative procedures in the areas to be treated within 3 months prior to initial treatment or plans for such treatment during the course of the Tixel2 device treatment, or before complete healing of such treatments has occurred.
* Any patient who takes or has taken any medications (including via topical application), herbal treatment (oral or topic), food supplements or vitamins, which may cause fragile skin or impaired skin healing during the last 3 months.
* Any patient who has used oral Isotretinoin (Accutane® or Roaccutan®) within 3 months prior to treatment or less.
* Any patient who has a history of bleeding coagulopathies or use of anticoagulants.
* Any patient who has tattoos or permanent makeup in the treated area.
* Any patient who has burned skin, blistered skin, irritated skin, or sensitive skin in any of the areas to be treated.
* Any patient who underwent thread lifting of the area to be treated in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-08-09 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
NIBUT in Seconds | 18 Weeks
  Non-Invasive Break Up Time
Ocular Surface Disease Index questionnaire | 18 Weeks
  Total 12 questions will be asked, ranked between 0-100. 0 being no dry eye symptoms and 100 severe dry eye symptoms.
SAFETY, number of AEs | 18 Weeks
  Any safety related event during the study will be recorded and analyzed

SECONDARY OUTCOMES:
Topography mm D | 18 Weeks
  Topography with K readings
Slit Lamp Exam; Normal, Abnormal | 18 Weeks
  Multiple Slit Lamp tests
Standardized Patient Evaluation of Eye Dryness (SPEED) Questionnaire | 18 Weeks
  Assessment of the frequency and severity of dry eye symptoms. scored 0 to 28; 0 being no dry eye symptoms and 28 severe dry eye symptoms.
Lid margin profile | 18 Weeks
  Lid margin profile
Tear Sampling Analysis | 18 Weeks
  ocular tear biomarkers
Staining; Total Ocular Staining Score | 18 Weeks
  Corneal staining fluorescein and conjunctival/lid margin staining lissamine green

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Shah, Phd, Principal Investigator — Midland Eye
Locations (1):
- Midland Eye, Solihull, United Kingdom

IPD SHARING:
Plan to Share IPD: No